CLINICAL TRIAL: NCT01629290
Title: In Vivo Comparison of Salivary Fluoride Levels Following the Application of Different 5% NaF Varnishes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Delta Dental Fund of Michigan (Other)
Responsible Party: Principal Investigator, Danika J Downey, Graduate Student, Restorative Dentistry, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00062943
Record Dates: First submitted 2012-06-10; First posted 2012-06-27 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Dental Cavity Lining

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Enamel Pro (Active Comparator): Varnish containing 5%NaF
  Interventions: Device: Enamel Pro
- Duraphat (Active Comparator): Varnish containing 5%NaF
  Interventions: Device: Duraphat
- Vanish (Active Comparator): Varnish containing 5%NaF
  Interventions: Device: Vanish
- Placebo (Placebo Comparator): Bland varnish containing no NaF
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Enamel Pro — Varnish treatment containing 5% NaF
  Other Names: Varnish
  Arms: Enamel Pro
Device: Duraphat — Varnish treatment containing 5% NaF
  Other Names: Varnish
  Arms: Duraphat
Device: Vanish — Varnish treatment containing 5% NaF
  Other Names: Varnish
  Arms: Vanish
Device: Placebo — Bland varnish containing no NaF
  Other Names: Bland varnish
  Arms: Placebo

SUMMARY:
This study will be a cross-over single blinded clinical study to evaluate the in vitro fluoride release of three different brands of 5% NaF varnish. The goal of this study is to determine if different formulations of varnish lead to differing amounts of fluoride release. Despite their similar concentrations of NaF (5%), some in vitro data have suggested that they may differ in the amount of fluoride release. Determining fluoride release of these varnishes in vivo is important in assessing both the safety and efficacy of the product.

DETAILED DESCRIPTION:
This study will be a cross-over single blinded clinical study to evaluate the in vitro fluoride release of three different brands of 5% NaF varnish. Subjects will be recruited at the University of Michigan School of Dentistry and will participate in a 15 minute clinical session at the beginning of each study arm, followed by 6 saliva collection recalls. During these sessions a fluoride varnish or placebo will be applied to their teeth, and subsequent salivary samples will be taken 1 hour, 4 hours, 6 hours, 24 hours, and 48 hours after the application. All subjects will receive 3 commercially available varnishes, and a placebo varnish. Between applications there will be a minimum of 2 weeks wash-out period. The goal of this study is to determine if different formulations of varnish lead to differing amounts of fluoride release. Despite their similar concentrations of NaF (5%), some in vitro data have suggested that they may differ in the amount of fluoride release. Determining fluoride release of these varnishes in vivo is important in assessing both the safety and efficacy of the product.

Specific Aims

1. Determine the concentration of fluoride available in the oral cavity at different time periods after the application of three different 5% NaF varnishes as measured in unstimulated human saliva.
2. Compare the different patterns of fluoride release from each of the varnishes by comparing the fluoride concentration in saliva at corresponding time periods .
3. Evaluate the validity of an in vitro model used to measure fluoride release from varnishes.

Percentage difference in fluoride release between the in vivo and in vitro data obtained from the same products will be compared. Because the comparison of different patterns of fluoride release from the varnishes is accomplished by analyzing the fluoride available concentration levels, it was an error to list that secondary aim as a secondary - or indeed any sort of outcome measure. The outcome measure data for "patterns of fluoride release" is exactly that which has been fully disclosed in the Primary Outcome Measure data tables. Therefore the secondary outcome measure previously listed: Compare the different patterns of fluoride release from each of the varnishes, which was really never properly an outcome measure, but an aim, has been deleted, with no loss of data transparency.

ELIGIBILITY:
Inclusion Criteria:

* All subjects between 18-65 years of age and do not fall under any of the exclusion criteria

Exclusion Criteria:

* Subjects with less than 20 teeth
* Subjects with significant untreated disease to include gum disease, extensive decay, or the need for pre-medication prior to dental treatment
* Pregnant or lactating women
* Subjects with a history of allergy to materials to be used in the study
* Subjects unable to produce adequate saliva for sampling
* Subjects deemed low risk for dental caries (no history of restorative work or presence of caries lesions)
* Subjects unable to be available for all 4 cycles of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Yaman, DDS, MS, Study Chair — University of Michigan; Gisele Neiva, DDS, MS, Study Chair — University of Michigan School of Dentsitry; Joseph Dennison, DDS, MS, Study Chair — University of Michigan; Carlos Gonzalez, DDS,MSD,PhD, Study Director — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Downey D, Dennison J, Eckert GJ, Flannagan SE, Neiva GF, Yaman P, Gonzalez-Cabezas C. Fluoride Levels in Unstimulated Whole Saliva following Clinical Application of Different 5% NaF Varnishes. Caries Res. 2018;52(6):431-438. doi: 10.1159/000485981. Epub 2018 Apr 3. PMID 29614502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 subjects were enrolled. All 15 subjects participated in the four arms/groups and received all four interventions for a total of 60 treatments.
Pre-assignment Details: Treatment consisted of the application of 0.4 ml of either a 5% NaF varnish, or a placebo (no fluoride) varnish applied to the buccal surfaces of all the teeth. After a minimum of 2 weeks washout period, the next randomly assigned treatment was given. All subjects received the 4 different treatments.
Groups:
- Varnishes and Placebo: Three dental varnishes with 5% NaF active ingredient (Enamel Pro, Duraphat and Vanish) and one bland varnish with no NaF applied to each subject at four timepoints.
  Each of the 15 participants received each of the four treatments, but the order followed was randomly arranged to be different, so there were twelve different patterns of assignment. Because all participants completed all four interventions, and the order was different for each, milestones are not used to indicate participation in each treatment, as that might imply a sequence, rather than simply that they received that intervention.
Period: Overall Study
Arm/Group | Varnishes and Placebo
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Varnish and Placebo: Three dental varnishes with 5% NaF active ingredient and placebo bland varnish containing no NaF
Arm/Group | Varnish and Placebo
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Fluoride Concentration and Release
Description: Fluoride release as measured by concentration of fluoride available in the oral cavity at different time periods after the application of 5% NaF varnish and placebo as measured in unstimulated human saliva
Time Frame: Baseline, 1 hr, 4 hrs, 6 hrs, 26 hrs and 50 hrs
Population: The 15 participants were each involved in each of the successive treatments with Enamel Pro, Duraphat, Vanish, and Placebo, (the order differed for each participant), and to show the differences between baseline and the different treatment levels, the baselines before each of the treatments is listed here along with the relevant treatment.
Measure: Mean (Standard Deviation); unit: ppm
Groups:
- Enamel Pro; Duraphat; Vanish: Dental varnish with 5% NaF active ingredient
Arm/Group | Enamel Pro | Duraphat | Vanish | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
ppm
  Baseline | .09 (.07) | .07 (.04) | .09 (.07) | .09 (.08)
  1 hr following application | 6.19 (4.09) | 18.94 (9.95) | 19.78 (14.57) | .02 (.02)
  4 hrs following application | .67 (.36) | 3.39 (4.83) | 4.12 (3.80) | .01 (.01)
  6 hrs following application | .37 (.2) | 1.82 (1.98) | 1.15 (.79) | .03 (.04)
  26 hrs following application | .4 (.02) | .19 (.15) | .2 (.33) | .02 (.04)
  50 hrs following application | .02 (.03) | .04 (.03) | .02 (.03) | .01 (.01)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Placebo: Placebo bland varnish containing no NaF
Arm/Group | Enamel Pro | Placebo | Duraphat | Vanish
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No